CLINICAL TRIAL: NCT02574702
Title: Prospective Randomized Controlled Trial to Reduce the Superficial Surgical Site Infection Due to a Contralateral Drainage Application in Loop Ileostomy Closure
Brief Title: Trial to Reduce Wound Infection With Contralateral Drainage in Loop Ileostomy Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Xavier Serra-Aracil, Medical Doctor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ILEOS-ISS_2013
Record Dates: First submitted 2013-03-18; First posted 2015-10-14 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Surgical Wound Infection
Keywords: superficial surgical site infection; loop ileostomy; Ileostomy closure
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Patients with primary loop ileostomy closure without drainage of the surgical wound
- Drainage Group (Experimental): Patients with the application of a contralateral drainage (Penrose ®) in surgical wound of primary loop ileostomy closure.
  Intervention: application of a contralateral drainage in surgical wound closure.
  Interventions: Procedure: application of a contralateral drainage (Penrose ® device)

INTERVENTIONS:
Procedure: application of a contralateral drainage (Penrose ® device) — application of a contralateral drainage (Penrose ®) in surgical wound of primary loop ileostomy closure
  Arms: Drainage Group

SUMMARY:
1. Introduction:

   The most common complication of loop ileostomies closure for rectal cancer patients undergoing a low anterior rectum resection, is the superficial surgical site infection (incidence 2-40%). There are various techniques related to closing loop ileostomy. In a retrospective study at our center, the investigators objectify that superficial surgical site infection rate was reduced by more than a half by the application of a contralateral drainage (Penrose ®) in primary loop ileostomy closure.
2. Objectives and Hypothesis:

   Hypothesis: The application of a contralateral drainage (Penrose ®) in primary loop ileostomy closure (in carriers of loop ileostomy by a low anterior rectum resection for rectal cancer) reduces the superficial surgical site infection.

   Main objective: To reduce the rate of superficial surgical site infection by the application of a contralateral drainage (Penrose ®) in surgical wound of primary loop ileostomy closure.
3. Methodology:

Prospective and randomized clinical trial on the effectiveness of contralateral Penrose® drainage implementation in those patients that have a primary loop ileostomy (by low anterior rectum resection) closure to be able to know if the investigators can reduce the superficial surgical site infection rate. Monitorization until 30 days after surgery

DETAILED DESCRIPTION:
1. Introduction:

   The most common complication of loop ileostomies closure for rectal cancer patients undergoing a low anterior rectum resection, is the superficial surgical site infection (incidence 2-40%). In the literature there are various techniques related to closing loop ileostomy that try to reduce the rate of infections recorded. In a retrospective study at our center, the investigators objectify that superficial surgical site infection rate was reduced by more than a half by the application of a contralateral drainage (Penrose ®) in primary loop ileostomy closure.
2. Objectives and Hypothesis:

   Hypothesis: The application of a contralateral drainage (Penrose ®) in primary loop ileostomy closure (in carriers of loop ileostomy by a low anterior rectum resection for rectal cancer) reduces the superficial surgical site infection.

   Main objective: To reduce the rate of superficial surgical site infection by the application of a contralateral drainage (Penrose ®) in surgical wound of primary loop ileostomy closure.

   Secondary objectives:
   * Identify risk factors associated with superficial surgical site infection in relation to a primary loop ileostomy closure (with or without drainage).
   * Reducing hospital stay and care at home.
3. Methodology:

Prospective and randomized clinical trial on the effectiveness of contralateral Penrose® drainage implementation in those patients that have a primary loop ileostomy (by low anterior rectum resection) closure to be able to know if the investigators can reduce the superficial surgical site infection rate.

It will be used a simple randomization. To assess the occurrence of superficial incisional infection, the investigators will be monitoring patients till 30 days after surgery

ELIGIBILITY:
Inclusion Criteria:

* Any patient carrying loop ileostomy due to low anterior resection for rectal cancer.
* Over 18 years.
* Surgery scheduled.
* Informed consent signed.

Exclusion Criteria:

Patients with terminal ileostomy.

* Patients with loop ileostomy different from any surgery of rectal cancer.
* To require another surgical procedure added.
* Urgent surgery.
* Patient refusal to participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with surgical site infection after ileostomy closure depending if there is or not a penrose drainage application | 30 days

SECONDARY OUTCOMES:
Number of patients with hematoma after ileostomy closure surgery | 30 days
Number of patients with seroma after ileostomy closure surgery | 30 days
Number of patients with anastomotic leak after ileostomy colsure surgery | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Serra-Aracil, MD, Principal Investigator — Hospital Universitario Parc Tauli de Sabadell
Locations (1):
- Hospital Universitario Parc Tauli de Sabadell, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Serracant A, Serra-Aracil X, Mora-Lopez L, Pallisera-Lloveras A, Serra-Pla S, Zarate-Pinedo A, Navarro-Soto S. The Effectiveness of Contralateral Drainage in Reducing Superficial Incisional Surgical Site Infection in Loop Ileostomy Closure: Prospective, Randomized Controlled Trial. World J Surg. 2019 Jul;43(7):1692-1699. doi: 10.1007/s00268-019-04972-6. PMID 30824960